CLINICAL TRIAL: NCT02242266
Title: A Single Dose, Placebo-controlled, Randomized, Double-blind, Double-dummy, Crossover Efficacy, Pharmacokinetics and Safety Comparison of Tiotropium Inhalation Powder (5 μg and 10 μg), Administered as the Bromide Salt From Hard Polyethylene Capsule Via the HandiHaler® 2 and Spiriva® HandiHaler® (18 μg Tiotropium) in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Pharmacokinetics and Safety Comparison of Tiotropium Inhalation Powder Administered as the Bromide Salt From Hard Polyethylene Capsule Via the HandiHaler® 2 and Spiriva® HandiHaler® in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1184.9
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

ARMS (4):
- Tiotropium low dose (Experimental): oral inhalation via the blue HandiHaler®
  Interventions: Drug: Tiotropium low dose; Drug: Placebo via the grey HandiHaler®
- Tiotropium medium dose (Experimental): oral inhalation via the blue HandiHaler®
  Interventions: Drug: Tiotropium medium dose; Drug: Placebo via the grey HandiHaler®
- Spiriva® HandiHaler® high dose (Active Comparator): oral inhalation via the grey HandiHaler®
  Interventions: Drug: Spiriva® HandiHaler® high dose; Drug: Placebo via the blue HandiHaler®
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo via the blue HandiHaler®; Drug: Placebo via the grey HandiHaler®

INTERVENTIONS:
Drug: Tiotropium low dose — inhalation powder, hard PE capsule
  Arms: Tiotropium low dose
Drug: Tiotropium medium dose — inhalation powder, hard PE capsule
  Arms: Tiotropium medium dose
Drug: Spiriva® HandiHaler® high dose — Tiotropium inhalation powder, hard gelatine capsule
  Arms: Spiriva® HandiHaler® high dose
Drug: Placebo via the blue HandiHaler® — oral inhalation via the blue HandiHaler®
  Arms: Placebo; Spiriva® HandiHaler® high dose
Drug: Placebo via the grey HandiHaler® — oral inhalation via the grey HandiHaler®
  Arms: Placebo; Tiotropium low dose; Tiotropium medium dose

SUMMARY:
The primary objective of this trial was to establish non-inferiority of lung function response to tiotropium 10 μg, formulated as inhalation powder in the polyethylene hard capsule and delivered via the HandiHaler® 2, compared to tiotropium 18 μg, formulated as inhalation powder in the hard gelatine capsule and delivered via the HandiHaler® (Spiriva®) following single dose inhalation in patients with COPD. A hard polyethylene (PE) capsule with half the strength (tiotropium 5 μg) was included to investigate a dose ordering effect.

The secondary objectives were to characterize the pharmacokinetics of tiotropium inhalation powder hard PE capsule (delivered via HandiHaler® 2) and tiotropium inhalation powder hard gelatine capsule (delivered via HandiHaler®) and to compare the safety of the two pharmaceutical formulations.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign an informed consent consistent with International Conference on Harmonization Good Clinical Practice (ICH-GCP) guidelines and local legislations prior to any study-related procedures, which includes medication washout and restrictions
2. All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria:

   Patients must have relatively stable* airway obstruction with a pre-dose FEV1 <= 60% of predicted normal and FEV1 <= 70% of FVC at Visits 1 and 2.
   * * The randomization of patients with any respiratory infection or COPD exacerbation in the 6 weeks prior to the Screening Visit (Visit 1) or during the baseline period should be postponed. Patients may be randomized 6 weeks following recovery from the infection or exacerbation
3. At Visit 1, patients must demonstrate an improvement in FEV1 of >= 12% over the baseline FEV1 value 45 minutes after inhalation of 4 puffs of 20 µg ipratropium bromide (Atrovent® MDI)
4. Male or female patients 40 years of age or older
5. Patients must be current or ex-smokers with a smoking history of more than 10 pack-years (Patients who had never smoked cigarettes had to be excluded)
6. Patients must be able to perform technically acceptable pulmonary function tests during the study period as required in the protocol
7. Patients must be able to inhale medication in a competent manner from the HandiHaler® 2 and the HandiHaler® devices

Exclusion Criteria:

1. Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
2. Patients with a recent history (i.e., six months or less) of myocardial infarction
3. Patients who have been hospitalized for heart failure (NYHA class III or IV) within the past year
4. Patients with any unstable or life threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year
5. Patients with malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years. Patients with treated basal cell carcinoma are allowed
6. Patients with a history of asthma, allergic rhinitis or atopy or who have a total blood eosinophil count ≥600/mm3. A repeat eosinophil count will not be conducted in these patients
7. Patients with a history of life threatening pulmonary obstruction, or a history of cystic fibrosis or clinically evident bronchiectasis
8. Patients with known active tuberculosis
9. Patients with significant alcohol or drug abuse within the past two years
10. Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criterion No. 1
11. Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the Screening Visit (Visit 1) or patients who are currently in a pulmonary rehabilitation program that will not be maintained throughout the duration of the study
12. Patients who regularly use daytime oxygen therapy for more than one hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy
13. Patients who are being treated with antihistamines (H1 receptor antagonists), antileukotrienes or leukotriene receptor antagonists for asthma or excluded allergic conditions. See exclusion criterion No 6
14. Patients who are being treated with cromolyn sodium or nedocromil sodium
15. Patients using oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day
16. Patients with known hypersensitivity to anticholinergic drugs, lactose or any other components of the inhalation capsule delivery system (Spiriva® HandiHaler®; tiotropium HandiHaler 2)
17. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception for the previous three months (i.e. oral contraceptives, intrauterine devices, diaphragm or subdermal implants, e.g.: Norplant®)
18. Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to Visit 1
19. Patients who have been treated with oral beta-adrenergics within one month prior to Visit 1 or during the run-in period
20. Patients who have been treated with theophylline preparations within one month prior to Visit 1 or during the run-in period
21. Patients who have been treated with the long-acting anticholinergic tiotropium (Spiriva®) within one month prior to Visit 1 or during the run-in period
22. Patients with any respiratory infections in the six weeks prior to the Screening Visit (Visit 1) or during the run-in period. In the case of a respiratory infection during the run-in period the latter may be extended up to six weeks
23. Patients who are currently participating in another study23. The randomisation of patients with any respiratory infection or COPD exacerbation in the six weeks prior to the Screening Visit (Visit 1) or during the baseline period should be postponed. Patients may be randomised six weeks following recovery from the infection or exacerbation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2005-07-28 (Actual); Primary Completion 2006-06-04 (Actual)

PRIMARY OUTCOMES:
Area under the curve for the time period 0 to 12 hours of forced expiratory volume in one second (FEV1 AUC0-12) | pre-dose and 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dosing

SECONDARY OUTCOMES:
Peak FEV1 on each test-day | pre-dose and 30, 60 minutes, 2 and 3 hours post-dosing
  Peak FEV1 is defined as the maximum FEV1 obtained within the first three hours post dosing
Peak forced vital capacity (FVC) | pre-dose and 30, 60 minutes, 2, 3, 4, 6, 8, 10, 12, 14, 22, 23 and 24 hours post-dosing
FVC AUC0-12 | pre-dose and 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dosing
FEV1 AUC12-24 | 12, 14, 22, 23 and 24 hours post-dosing
FEV1 AUC0-24 | pre-dose and 30, 60 minutes, 2, 3, 4, 6, 8, 10, 12, 14, 22, 23 and 24 hours post-dosing
FVC AUC12-24 | 12, 14, 22, 23 and 24 hours post-dosing
FVC AUC0-24 | pre-dose and 30, 60 minutes, 2, 3, 4, 6, 8, 10, 12, 14, 22, 23 and 24 hours post-dosing
Individual FEV1 measurements at each time point | pre-dose and 30, 60 minutes, 2, 3, 4, 6, 8, 10, 12, 14, 22, 23 and 24 hours post-dosing
Individual FVC measurements at each time point | pre-dose and 30, 60 minutes, 2, 3, 4, 6, 8, 10, 12, 14, 22, 23 and 24 hours post-dosing
AUCt1-t2 (area under the concentration-time curve of the analyte in plasma over the time interval t1 to t2) | 5, 15, 30 minutes, 1 and 2 hours following drug administration
Cmax (maximum measured concentration of the analyte in plasma) | 5, 15, 30 minutes, 1 and 2 hours following drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | 5, 15, 30 minutes, 1 and 2 hours following drug administration
Aet1-t2 (amount of analyte that is eliminated in urine from the time point t1 to time point t2) | 0 to 2, 2 to 12 hours after administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | 0 to 2, 2 to 12 hours after administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | 0 to 2, 2 to 12 hours after administration
%AUCtz-∞ (percentage of the extrapolated part of the total AUC0-∞) | 5, 15, 30 minutes, 1 and 2 hours following drug administration
Number of patients with adverse events | up to 13 weeks